CLINICAL TRIAL: NCT03678844
Title: Effect of Taekwondo Practice on Cognitive Function in Adolescents With Attention Deficit Hyperactivity Disorder
Brief Title: Taekwondo Practice in Adolescents With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Maamer Slimani, Principal Investigator, University of Genova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TKD0012
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taekwondo practice (Experimental)
  Interventions: Behavioral: Taekwondo practice; Other: CONTROL
- CONTROL (Placebo Comparator)
  Interventions: Behavioral: Taekwondo practice; Other: CONTROL

INTERVENTIONS:
Behavioral: Taekwondo practice — The Taekwondo intervention program consisted of the technical skill development aspect (e.g., blocking, punching and kicking) of the sport and poomse (forms) for 30-min.
Other: CONTROL — The participants of the control group engaged in physical activities, including athletics, handball and gymnastic, during two sessions of physical education per week at school.

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is one of the most common neuro-developmental/behavioral disorders among adolescents. Sport and physical activity seem to play a major role in the development of cognition, memory, selective attention and motor reaction time, especially among adolescents with ADHD. In this context, the objective of this study was to investigate the effects of a one and a half year long Taekwondo (TKD) intervention on cognitive function in adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with Attention Deficit Hyperactivity Disorder

Exclusion Criteria:

* Participants with good attentional performance

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Stroop | 45 seconds
  Participants are presented with a page consisting of five columns, each with 20 items for a total of 100 items per page.

SECONDARY OUTCOMES:
Ruff 2 and 7 | 5 minutes
  This test consists of a series of 20 blocks (10 blocks of digits only and 10 blocks of both digits and letters).

IPD SHARING:
Plan to Share IPD: No
Overall data